CLINICAL TRIAL: NCT01455727
Title: Pharmaceutical Care of Ambulatory Elderly Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantou Hospital (Other Government)
Responsible Party: Principal Investigator, Jyun-Hong Chen, Clinical Pharmacist, Pharmacy Department, Nantou Hospital, Nantou Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 100B4022-100MID-08
Record Dates: First submitted 2011-10-14; First posted 2011-10-20 (Estimated); Last update posted 2012-09-17 (Estimated); Status verified 2012-09

CONDITIONS: Diabetes Mellitus
Keywords: Pharmaceutical care; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Pharmaceutical Services

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Pharmaceutical care (Experimental): The Pharmacist provided Pharmaceutical care on the ambulatory elderly Diabetes patients, provided recommendation to the physician and reffered the patients to other diabetes-care-team members, including the CDEs and dietitians.
  Interventions: Other: Pharmaceutical care
- Usual care (Active Comparator): Patients received usual care directed by their physician.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Pharmaceutical care — The Pharmacist provided Pharmaceutical care on the ambulatory elderly Diabetes patients, provided recommendation to the physician and reffered the patients to other diabetes-care-team members, including the CDEs and dietitians.
  Arms: Pharmaceutical care
Other: Usual care — Control patients received usual care directed by their physician.
  Arms: Usual care

SUMMARY:
This trial will try to perform pharmaceutical care on ambulatory elderly diabetes patients. To provide appropriate diabetes education administration, identify and resolve drug-related problems, assess the appropriateness of their medications, establish the mechanism of medication consultations. Each patient will be assessed by the MMSE(Mini-Mental State Examination) and GDS(Geriatric Depression Scale). The effectiveness of pharmacist's intervention will be assessed by lab data and some questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older
* A1c greater than or equal to 9.0

Exclusion Criteria:

* Not expected to live for the duration of the study
* Unwillingness to participate and attend pharmacist visits
* Unwillingness to participate the questionnaires(MMSE, GDS)

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Hgb A1c change | 12 month
  baseline, second measurement during 3 to 6 month after baseline, and the last measurement during 9 to 12 month after baseline

SECONDARY OUTCOMES:
Mini-Mental State Examination(MMSE) Score change | 1 year
  baseline and the second test was performed after 3 month.
Taiwan Geriatric Depression Scale(GDS) Score change | 1 year
  baseline and the second test was performed after 3 month.

CONTACTS AND LOCATIONS:
Locations (1):
- Nantou Hospital, Nantou City, Taiwan